CLINICAL TRIAL: NCT04348331
Title: Magnetic Resonance Imaging Pulse Sequences in Diagnosis of Temporomandibular Disorders
Brief Title: Dual-echo and Inversion Recovery Magnetic Resonance Imaging Pulse Sequences in Diagnosis of Temporomandibular Disorders. Diagnostic Accuracy Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Khalifa Zayet, Professor Oral and Maxillofacial Radiology, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: ORAD 7:1:1
Record Dates: First submitted 2020-04-09; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Dual echo MRI sequence — new MRI sequences for imaging of joints
  Other Names: Fluid-attenuated inversion recovery (FLAIR) MRI sequence; Short-TI Inversion Recovery (STIR) MRI sequence

SUMMARY:
In the present study, investigators are going to investigate the potential of inversion recovery (fluid attenuated inversion recovery -FLAIR and short-TI Inversion Recovery -STIR) sequence images to demonstrate joint effusion, compared to T2-weighted images.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pain related to temporomandibular joint.
* Patients with limited mouth opening.

Exclusion Criteria:

* Patients with pain related to temporomandibular joint for less than one month duration.
* Patients with limited mouth opening for less than one month duration.
* Patients with history of TMJ surgical intervention.
* Patients with history of TMJ arthrocentesis.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Identification of temporomandibular joint effusion. | through study completion, an average of 1 year
  Binary outcome measure

SECONDARY OUTCOMES:
Delineation of temporomandibular joint disc position. | through study completion, an average of 1 year
  Descriptive measure: 10 - 12 - 2 o'clock position

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed K Zayet, Study Director — Cairo University
Locations (1):
- Nouran Nabil Marzaban, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No